CLINICAL TRIAL: NCT05925543
Title: Outcome of Kasai Portoenterostomy in Biliary Atresia in Upper Egypt
Status: Completed | Type: Observational
Sponsor: Aswan University Hospital (Other)
Responsible Party: Principal Investigator, Sarah Magdy Abdelmohsen, Lecturer, Aswan University Hospital
Other Study IDs: Aswan UH7
Record Dates: First submitted 2023-06-22; First posted 2023-06-29 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Biliary Atresia
Keywords: Cholestasis; Neonate jaundice; Cholangitis; Short-term outcome; Survival with the native liver
MeSH Terms: conditions — Biliary Atresia; Cholestasis; Cholangitis

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- all neonates diagnosed with biliary atresia and managed by Kasai portoenterostomy.: all neonates diagnosed with biliary atresia in the previous period 2019 and managed by Kasai portoenterostomy.
  Interventions: Procedure: Kasai portoenterostomy operation.

INTERVENTIONS:
Procedure: Kasai portoenterostomy operation. — Kasai portoenterostomy operation for biliary atresia patients.
  Other Names: Kasai operation

SUMMARY:
Kasai portoenterostomy is the key standard operation for biliary atresia. The aim of the study is to evaluate the short-term outcome of Kasai portoenterostomy for biliary atresia infants in Upper Egypt.

DETAILED DESCRIPTION:
It is a cross-sectional retrospective multicenter study from Upper Egypt. The data will collected from the medical records of three university hospitals in Upper Egypt from January 2019 to December 2019.

Inclusion and exclusion criteria

Inclusion criteria included all neonates diagnosed with biliary atresia in the previous period and managed by Kasai portoenterostomy.

Exclusion criteria were neonates without a confirmed diagnosis of biliary atresia.

ELIGIBILITY:
Inclusion Criteria:

* all neonates diagnosed with biliary atresia in the previous period and managed by Kasai portoenterostomy.

Exclusion Criteria:

* Exclusion criteria were neonates without a confirmed diagnosis of biliary atresia.

Ages: 4 Weeks to 19 Weeks | Sex: All
Age Groups: Child
Study Population: all neonates diagnosed with biliary atresia in the previous period (2019) and managed by Kasai portoenterostomy.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
the rate of jaundice clearance | from 3 months up to one year
  the clearance of jaundice measured by total serum bilirubin < 1.2 mg \ dL and direct bilirubin < 0.3 mg dL within one year postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Abdelmohsen, Md, Principal Investigator — Aswan University Hospital
Locations (1):
- Aswan university Hospital, Aswān, Aswan Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
It was a cross-sectional retrospective multicenter study from Upper Egypt. The data will collect from the medical records of three university hospitals in Upper Egypt from January 2019 to December 2019.
Supporting Information: Study Protocol
Time Frame: January 2019- December 2019
Access Criteria: Biliary Atresia in Upper Egypt